CLINICAL TRIAL: NCT00085098
Title: Radiotherapy Alone Versus Chemotherapy Followed By Response-Based Radiotherapy For Newly Diagnosed Primary CNS Germinoma
Brief Title: Radiation Therapy Compared With Chemotherapy and Radiation Therapy in Treating Patients With Newly Diagnosed Primary Central Nervous System (CNS) Germ Cell Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0232; CDR0000367294 (Other: Clinical Trials.gov); COG-ACNS0232 (Other: Children's Oncology Group)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2013-11-06 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Brain Tumor; Central Nervous System Tumor
Keywords: childhood central nervous system germ cell tumor
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; etoposide phosphate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (radiotherapy only) (Experimental): Within 52 days of surgery, patients will undergo standard-dose radiation therapy 5 days a week for approximately 5-6 weeks.
  Interventions: Radiation: radiation therapy
- Regimen B (chemotherapy plus radiotherapy) (Experimental): Courses 1 and 2: Patients receive carboplatin IV over 1 hour on days 1 and 2 and etoposide IV over 2 hours on days 1-3. Treatment repeats every 21 days for 2 courses.
  Within 3 weeks of completing chemotherapy, patients with CR undergo low-dose radiation therapy 5 days a week for 5 weeks. Patients with MRD, a PR, or SD receive chemotherapy courses 3 and 4 as outlined below.
  Courses 3 and 4: Patients receive cisplatin IV over 6 hours on day 1, cyclophosphamide IV over 1 hour on days 2 and 3, and filgrastim (G-CSF), subcutaneous (SC) or IV beginning on day 4 and continuing until blood counts recover.
  Treatment repeats every 21 days for 2 courses. Patients achieving a CR or MRD proceed to reduced-dose radiotherapy. Patients with a PR, SD, or progressive disease (PD) are restaged and may undergo standard radiation therapy as in regimen A. Reduced-dose radiation therapy: Within 6 weeks of starting course 4, patients undergo lower-dose radiation therapy once daily on days 1-5 for 5 weeks
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given by infusion or injection
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #61462
  Arms: Regimen B (chemotherapy plus radiotherapy)
Drug: carboplatin — Given IV over 1 hour
  Other Names: Paraplatin; NSC #241240
  Arms: Regimen B (chemotherapy plus radiotherapy)
Drug: cisplatin — Given IV over 6 hours
  Other Names: Cis-diamminedichloroplatinum II; Platinol-AQ; NSC #119875
  Arms: Regimen B (chemotherapy plus radiotherapy)
Drug: cyclophosphamide — Given IV over 1 hour
  Other Names: Cytoxan; NSC #26271
  Arms: Regimen B (chemotherapy plus radiotherapy)
Drug: etoposide — Given IV over 2 hours
  Other Names: VePesid; Etopophos; VP-16; NSC #141540
  Arms: Regimen B (chemotherapy plus radiotherapy)
Radiation: radiation therapy — Patients undergo radiotherapy 5 days a week

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether radiation therapy alone is as effective as chemotherapy plus radiation therapy in treating germ cell tumor.

PURPOSE: This randomized phase III trial is studying radiation therapy alone to see how well it works compared to chemotherapy and radiation therapy in treating patients with newly diagnosed primary CNS germ cell tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare event-free survival and overall survival of patients with newly diagnosed primary CNS germ cell tumor treated with conventional radiotherapy alone (regimen A) vs chemotherapy followed by tumor response-based radiotherapy (regimen B).

Secondary

* Determine the complete response rate in patients treated with regimen B.
* Determine the acute and subacute toxicity of regimen B in these patients.
* Compare treatment-related morbidity, in terms of verbal learning and memory, executive functioning, and quality of life, in patients treated with these regimens.
* Determine the prognostic value of baseline serum, lumbar, and intraventricular levels of human chorionic gonadotropin levels from patients treated with these regimens.
* Determine the prognostic value of extent of disease (M+ vs modified M+ vs M0) on event-free survival and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor location (pineal vs suprasellar vs pineal + suprasellar or other), and disease stage (disseminated vs occult multi-focal vs localized). Patients are randomized to 1 of 2 treatment regimens.

All patients undergo an operative procedure (endoscopic biopsy, stereotactic biopsy, or open craniotomy) to confirm the diagnosis of pure germ cell germinoma followed by an intraoperative and perioperative staging evaluation.

* Regimen A (radiotherapy only): Within 52 days of surgery, patients undergo standard-dose radiotherapy once daily on days 1-5 for approximately 5-6 weeks.
* Regimen B (chemotherapy plus radiotherapy):

  * Courses 1 and 2: Patients receive carboplatin IV over 1 hour on days 1 and 2 and etoposide IV over 2 hours on days 1-3. Treatment repeats every 21 days for 2 courses.

Patients achieving a complete response (CR) proceed to reduced-dose radiotherapy. Patients with minimal residual disease (MRD), a partial response (PR), or stable disease (SD) receive chemotherapy courses 3 and 4 as outlined below. Patients with progressive disease undergo a second surgical procedure for biopsy and are restaged. Patients with a confirmed diagnosis of germ cell tumor with no change in tumor markers and no new lesions after restaging proceed to chemotherapy courses 3 and 4.

* Courses 3 and 4: Patients receive cisplatin IV over 6 hours on day 1, cyclophosphamide IV over 1 hour on days 2 and 3, and filgrastim (G-CSF) subcutaneously or IV beginning on day 4 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses.

Patients achieving a CR or MRD proceed to reduced-dose radiotherapy. Patients with a PR, SD, or progressive disease are restaged. Patients with a confirmed diagnosis of germ cell tumor after restaging undergo standard radiotherapy as in regimen A.

* Reduced-dose radiotherapy: Within 6 weeks of starting course 4, patients undergo lower-dose radiotherapy once daily on days 1-5 for 5 weeks.

Treatment in both regimens continues in the absence of unacceptable toxicity or in the event that a non-germinomatous germ cell tumor is detected.

Quality of life and neuropsychological function within the domains of intelligence, attention-concentration, memory, and executive functioning are assessed at 9, 30, and 60 months after diagnosis.

Patients are followed every 4 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 225 patients (approximately 112 per treatment regimen) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS pure germ cell tumor

  * Diagnosed within the past 31 days
* Meets any 1 OR none (i.e., M0 [localized disease]) of the following staging criteria:

  * M+ (disseminated disease)

    * Leptomeningeal or intraventricular metastases visualized on MRI scans of the brain and spine
    * Clumps of tumor cells on lumbar cerebrospinal fluid (CSF) cytology
    * Visible tumor studding the walls of the lateral or third ventricles noted during endoscopy or surgery
    * Primary tumor arising within the parenchyma of the brain, brainstem, or spinal cord
    * Measurable multi-focal tumors arising in both the pineal and suprasellar regions (i.e., multiple midline tumors)
    * Infiltrative, intra-axial extension on brain MRI > 1 cm beyond enhancing tumor
  * Modified M+ (occult multi-focal disease)

    * M0 at diagnosis with a localized pineal region tumor with signs and symptoms of diabetes insipidus without measurable disease in the suprasellar region
* Lumbar CSF assay meeting criteria for the following marker profiles:

  * Serum and CSF beta human chorionic gonadotropin (β-HCG) ≤ 50 IU/dL
  * Serum alpha fetoprotein (AFP) ≤ 10 IU/L AND ≤ institutional norm
  * CSF AFP ≤ 2.0 IU/L AND ≤ institutional norm

PATIENT CHARACTERISTICS:

Age

* 3 to 25

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3 (transfusion independent)
* Hemoglobin > 10.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 times ULN

Renal

* Creatinine adjusted according to age as follows*:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male]) AND
* Creatinine clearance OR radioisotope glomerular filtration rate > 70 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Euthyroid (with or without levothyroxine sodium therapy) as determined by normal T4 ± thyroid-stimulating hormone levels*
* Diabetes insipidus allowed provided patient is relatively stable on desmopressin acetate
* Normal endogenous cortisol function*
* Adequate antidiuretic hormone reserves* NOTE: *Unless receiving replacement therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent replacement hormones allowed (e.g., corticosteroids, levothyroxine sodium, and desmopressin acetate)

Radiotherapy

* Not specified

Surgery

* Prior surgery for germ cell tumor allowed

Other

* No other prior therapy for germ cell tumor
* Concurrent anticonvulsants allowed

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C. Allen, MD, Study Chair — NYU Langone Health
Locations (107):
- United States (95):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Sutter Cancer Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (8):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
- San Jorge Children's Hospital, Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen B (Chemotherapy Plus Radiotherapy): Courses 1,2:Patients (PTS) receive carboplatin IV over 1 hour on days 1-2 and etoposide IV over 2 hours on days 1-3. Treatment repeats every 21 days for 2 courses. Within 3 weeks of completing chemotherapy, PTS with complete response (CR) undergo low-dose radiation therapy 5 days a week for 5 weeks. PTS with minimal residual disease (MRD), a PR, or stable disease (SD) receive chemotherapy courses 3,4. Courses 3,4:PTS receive cisplatin IV over 6 hours on day 1, cyclophosphamide IV over 1 hour on days 2-3 and filgrastim (G-CSF) subcutaneous (SC) or IV on day 4 continuing until blood counts recover. Treatment repeats every 21 days for 2 courses. PTS achieving a CR or MRD proceed to reduced-dose radiotherapy. PTS with a partial response (PR), SD or progressive disease (PD) are restaged and may undergo standard radiation therapy as in regimen A.Reduced-dose radiation therapy: Within 6 weeks of starting course 4, PTS undergo lower-dose radiation therapy once daily on days 1-5 for 5 weeks.
Period: Overall Study
Arm/Group | Regimen A (Radiotherapy Only) | Regimen B (Chemotherapy Plus Radiotherapy)
Started | 11 | 13
Completed | 10 | 11
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligible | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Regimen B (Chemotherapy Plus Radiotherapy): Courses 1 and 2: Patients receive carboplatin IV over 1 hour on days 1 and 2 and etoposide IV over 2 hours on days 1-3. Treatment repeats every 21 days for 2 courses.
  Within 3 weeks of completing chemotherapy, patients with CR undergo low-dose radiation therapy 5 days a week for 5 weeks. Patients with MRD, a PR, or SD receive chemotherapy courses 3 and 4 as outlined below.
  Courses 3 and 4: Patients receive cisplatin IV over 6 hours on day 1, cyclophosphamide IV over 1 hour on days 2 and 3, and filgrastim (G-CSF) SC or IV beginning on day 4 and continuing until blood counts recover.
  Treatment repeats every 21 days for 2 courses. Patients achieving a CR or MRD proceed to reduced-dose radiotherapy. Patients with a PR, SD, or PD are restaged and may undergo standard radiation therapy as in regimen A.
  Reduced-dose radiation therapy: Within 6 weeks of starting course 4, patients undergo lower-dose radiation therapy once daily on days 1-5 for 5 weeks
- Total: Total of all reporting groups
Arm/Group | Regimen A (Radiotherapy Only) | Regimen B (Chemotherapy Plus Radiotherapy) | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 13 | 23
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18
  Australia | 1 | 4 | 5
  Switzerland | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Data will be summarized as number of patients in the following categories at the time of data cutoff for analyses of 3-year EFS: 1)Experienced a qualifying event (QE) (see below);2)Event-free through 3 years of follow-up;3)Event-free until data cutoff (if less than 3 years of follow-up);4)Withdrew from study;5)Lost to follow-up.
  QEs: 1)disease progression, defined as increase >= 40% in tumor volume or >= 25% in tumor area of target lesions;2)development of new lesions;3)occurrence of a second malignant neoplasm, defined as a malignancy with different histological type from trial-qualifying diagnosis;4)death from any cause.
  Stat. analyses will be based on time from enrollment to the earliest of: 1)occurrence of any of the QEs;2)withdrawal from study or lost to follow-up;3)completion of three years of follow-up event-free;4)data cutoff for completion of the statistical analyses for the protocol's primary objective.
  NOTE: Reported data are through May 2009 (see Caveats section).
Time Frame: Study enrollment until date of earliest qualifying event (QE), date last known to be QE-free if the patient is followed for less than three years and is QE-free at the time of analysis, or 3 years if the patient is QE-free at 3 years
Population: By protocol design, all eligible patients were considered in the evaluation of primary study aim. Two (2) patients were considered ineligible. All other patients (10 enrolled to regimen A and 12 enrolled to regimen B) are included in the evaluation for the primary outcome measure.
Measure: Number; unit: participants
Arm/Group | Regimen A (Radiotherapy Only) | Regimen B (Chemotherapy Plus Radiotherapy)
Number analyzed (Participants) | 10 | 12
participants
  Experienced a qualifying event | 1 [43 to 98] | 1 [54 to 99]
  Event-free through 3 years of follow-up | 0 | 0
  Event-free at data cutoff (if < 3 years follow-up) | 9 | 11
  Withdrew from study prior to 3 years of follow-up | 0 | 0
  Lost to follow-up prior to 3 years of follow-up | 0 | 0

2. Secondary Outcome: Number of Participants With a Response to Regimen B
Description: To assess the complete response rate to pre-radiotherapy chemotherapy (Reg B only). Response was determined after completing 2-4 cycles of chemotherapy on Reg B. Complete Response (CR) is defined as disappearance of all target lesions.
Time Frame: 5 years from beginning of treatment
Population: Patients who were treated in Regimen B and had at least one response assessment are included in this analysis. One patient in Regimen B withdrew from the pre-Radiotherapy chemotherapy and did not have any response assessment were not included for the response analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen B (Chemotherapy Plus Radiotherapy)
Number analyzed (Participants) | 11
Participants | 8

3. Secondary Outcome: Toxicity and Safety as Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: The analysis of toxicity will focus on estimating the rates of key acute and subacute toxicity occurring during the first induction chemotherapy. The list of toxicities of interest include Anemia or Febrile Neutropenia; Nausea or Vomiting; Infections and Infestations; Neutrophil or White blood count decrease; and Hypokalemia or Hyponatremia
Time Frame: From the beginning of treatment, assessed up to 5 years
Population: Patients who received any pre-radiotherapy chemotherapy in Regimen B
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen B (Chemotherapy Plus Radiotherapy)
Number analyzed (Participants) | 12
Participants
  Anemia or Febrile Neutropenia | 2
  Nausea or Vomiting | 2
  Infections and Infestations | 2
  Neutorphil or White blood count decrease | 7
  Hypokalemia or Hyponatremia | 3

4. Secondary Outcome: Quality of Life (QOL) and Neurocognitive Assessment (NP)
Description: The primary endpoints for QOL and NP assessments will be the global scale value from each of these instruments at the two-year time point. Analyses of subscales (if they exist) and of assessments at other times will be of secondary interest. It is assumed that scale values are standardized to a reference normal population. The scores range from 0 to 100 with higher score reflecting better QoL or neurocognitive assessment.
Time Frame: 2 years from beginning of treatment
Population: All eligible patients who also successfully completed therapy and were assessed for quality of life and neurocognitive outcome.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Regimen A (Radiotherapy Only) | Regimen B (Chemotherapy Plus Radiotherapy)
Number analyzed (Participants) | 10 | 11
Scores on a scale
  Overall IQ Score: number analyzed (Participants) | 5 | 7
  Overall IQ Score | 98.60 (17.95) | 92.43 (6.27)
  Self Report Score-Internalizing Problems: number analyzed (Participants) | 2 | 4
  Self Report Score-Internalizing Problems | 41.00 (2.83) | 42.50 (5.51)
  Self Report Score-Emotional Problems: number analyzed (Participants) | 2 | 4
  Self Report Score-Emotional Problems | 44.00 (2.83) | 42.00 (4.55)
  Self Report Score-Personal Adjustment Strengths: number analyzed (Participants) | 2 | 4
  Self Report Score-Personal Adjustment Strengths | 51.50 (2.12) | 60.50 (3.32)
  Parent Report QoL Total Score: number analyzed (Participants) | 2 | 2
  Parent Report QoL Total Score | 88.04 (6.15) | 79.35 (6.15)
  Self Report QoL Total Score: number analyzed (Participants) | 1 | 2
  Self Report QoL Total Score | 95.65 (NA) — The Reg A only has 1 pt with Self Report QoL Total Score, so the Standard Deviation cannot be estimated. | 90.76 (0.76)

ADVERSE EVENTS:
Time Frame: During protocol therapy; six months (maximum).
Description: All eligible patients were considered in the evaluation of adverse events (AEs). Two patients were considered ineligible. All other patients (10 enrolled to regimen A and 12 enrolled to regimen B) are included in AE reporting.
  Systematic assessment was performed according to protocol-directed schedule of assessments, and as clinically indicated.
Arm/Group | Regimen A (Radiotherapy Only) | Regimen B (Chemotherapy Plus Radiotherapy)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 4/10 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Radiotherapy Only) (N=10) | Regimen B (Chemotherapy Plus Radiotherapy) (N=12)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
"Infections and infestations - Other, specify" (Infections and infestations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
"Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify" (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 9 (9)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 7 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
Study closed early due to slow accrual. Analysis plans were not carried out (lack of statistical precision compromised the ability to draw appropriate conclusions). Reported Primary Outcome Measure data reflects data collection through May 2009.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No